CLINICAL TRIAL: NCT01699672
Title: Cancer Patients' Knowledge and Satisfaction After Group-based or Individual Information About Their Disease and Treatment Plan
Brief Title: Group-based or Individual Information About Disease and Treatment Plan
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Problems recruiting patients (not willing, travel time, no respons)
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REK2012/1238
Record Dates: First submitted 2012-09-21; First posted 2012-10-04 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Prostate Cancer; Breast Cancer
Keywords: Patient education; information; communication
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group and Individual information (Experimental): The patients will receive two 1.5-2 hour standardized validated group information sessions in addition to regular information from their doctors and nurses.
  Interventions: Other: Group information
- Individual information (No Intervention): Standard information about disease and treatment from doctor and nurse given at 2 occasions.

INTERVENTIONS:
Other: Group information — The patients will receive two 1.5-2 hour standardized validated group information sessions in addition to regular information from their doctors and nurses.
  Arms: Group and Individual information

SUMMARY:
The main aim of the current study is to investigate whether the addition of a standardized,group-based educational program to the information provided by health care personnel improves cancer patients' knowledge level about their disease, planned treatment and common side-effects of the treatment.

Secondary aims are to investigate if the addition of the educational program increases the likelihood of completing treatment as planned, reduces level of anxiety, reduces the frequency of serious side effects, increases patient reported health related quality of life, and increases the degree of patient satisfaction with respect to how they have received the information before, during and after treatment.

DETAILED DESCRIPTION:
There are strong indications that group-based information provides better information for cancer patients about their disease, treatment options - and potential benefits and side effects of the planned therapy than information provided during a regular doctor consultation.

The investigators believe that standardizing and repeating the information as well as having more time for questions in an open environment for reflections will improve the amount of information patients can perceive. Furthermore, all patients will be given written information.

Better-informed patients may be more motivated and may contact health care personnel earlier than other patients when they develop side effects. This may reduce the risk of serious treatment-related complications and increase the chances of patients completing the planned treatment. But none have compared to what extent an organization like Vardesenteret improves the patients' knowledge and whether patients are more satisfied with these methods for informing them. Results from studies on the influence of patient anxiety and distress on patient's abilities to perceive information are conflicting.Two large groups of relatively homogenous cancer patients are patients with lower-stage breast cancer patients who are eligible for adjuvant chemotherapy and patients with localized prostate cancer eligible for curative radiotherapy.

ELIGIBILITY:
Inclusion criteria:

* Breast cancer patients that are candidates for adjuvant chemotherapy after surgery.
* Prostate cancer patients that are candidates for curative radiotherapy
* Signed informed consent
* Patient expected to be able to complete the planned treatment and the study procedures
* 18years or older

Exclusion Criteria:

-Patients not fulfilling inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Knowledge | 1 week
  Knowledge questionnaires specially made for the study. Constructed as statements with response categories; correct, false and don´t know.
Knowledge | 2 weeks
  Knowledge questionnaires specially made for the study. Constructed as statements with response categories; correct, false and don´t know.
Knowledge | 9 weeks
  Knowledge questionnaires specially made for the study. Constructed as statements with response categories; correct, false and don´t know.

SECONDARY OUTCOMES:
Quality of Life | 9 weeks
  European Organization for Research and Treatment of Cancer Core Quality-of-Life Questionnaire C30
Patients Subjective state of information | 1 week
  European Organization for Research and Treatment of Cancer Core Quality-of-Life Questionnaire INFO 25
Patients Subjective state of information | 2 weeks
  European Organization for Research and Treatment of Cancer Core Quality-of-Life Questionnaire INFO 25
Patients Subjective state of information | 9 weeks
  European Organization for Research and Treatment of Cancer Core Quality-of-Life Questionnaire INFO 25
Anxiety | 1 week
  STAI-State and Trait Anxiety Inventory
Anxiety | 2 weeks
  STAI-State and Trait Anxiety Inventory
Anxiety | 9 weeks
  STAI-State and Trait Anxiety Inventory
Adverse events | 2 weeks
  CTCEA, Common Terminology Criteria for Adverse Events
Adverse events | 9 weeks
  CTCEA, Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Stein Kaasa, MD, Prof., Principal Investigator — St Olavs Hospital - Trondheim University Hospital and PRC, European Palliative Care Research Center; Ola Berger, MD, Study Director — St Olavs Hospital - Trondheim University Hospital and PRC, European Palliative Care Research Center; Bjørn H Gønberg, MD, PhD, Study Chair — St Olavs Hospital - Trondheim University Hospital and PRC, European Palliative Care Research Center; Kari Sand, Cand Philol, Study Chair — PRC, European Palliative Care Research Center; Jo Å Lund, MD, PhD, Study Chair — St Olavs Hospital - Trondheim University Hospital and PRC, European Palliative Care Research Center; Jon H Loge, MD, Prof., Study Chair — National Resource Centre for Studies of Late Effects after Cancer Treatment, Oslo University Hospital, Radiumhospitalet, Oslo, Norway; Department of Behavioral Sciences in Medicine, University of Oslo
Locations (1):
- St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Derived] Berger O, Gronberg BH, Loge JH, Kaasa S, Sand K. Cancer patients' knowledge about their disease and treatment before, during and after treatment: a prospective, longitudinal study. BMC Cancer. 2018 Apr 3;18(1):381. doi: 10.1186/s12885-018-4164-5. PMID 29614997